CLINICAL TRIAL: NCT00904956
Title: Study of Latent Tuberculosis Infection (LTBI) by High Resolution Scanner
Acronym: GRANLATHU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: CIBERES CRP-TB program (Unknown)
Responsible Party: Pere-Joan Cardona, Fundació Institut Germans Trias i Pujol
Other Study IDs: GRANLATHU
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2009-11

CONDITIONS: Tuberculosis
Keywords: Latent Tuberculosis Infection; High Resolution Scanners; Dynamic Hypothesis of Latent Tuberculosis Infection
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
It is traditionally considered that someone with a positive tuberculin skin test (TST) (and/or positive result in Cell Interferon-Gamma Release Assay (TIGRA), depending on the different countries' guidelines) is infected but not ill when the absence of lesions is demonstrated in a thorax X-Ray assay. Even though, the experiences described in literature using cows and pigs as animal models for the study of LTBI demonstrate the presence of this kind of lesion in the animals, even too small to be detected by X-Ray assay, which would suggest they also could happen in human LTBI. Nowadays, the High Resolution Scanners (HR TC) offer the possibility of detecting any lesion approximately 1 mm in diameter, so the investigators plan to use this technique to screen people already infected by M. tuberculosis (but not ill, following the Diagnosis Standard Guidelines).

Additional pathological analysis of resected and post-mortem tissues will provide lesion-based profiles of humans infected with tuberculosis.

DETAILED DESCRIPTION:
It is traditionally considered that the development of LTBI is due to the M. tuberculosis ability to develop a dormancy state within well-structured lesions (granulomas), which can remain in the lung of the host even for life. The investigators have developed a new original hypothesis based on scientific evidence that takes into account the idea that a lesion cannot be held forever, because the host tends to remove any lesion in order to rebuild the original parenchyma, in a healing process. Even if M. tuberculosis can remain in a dormant/non-replicating state for a long period, this is an important but not sufficient factor to explain the LTBI. The Dynamic Hypothesis tries to explain the existence of LTBI in spite of the healing process that could remove it by a constant reinfection of the host's tissue.

ELIGIBILITY:
Inclusion Criteria:

* People with TST+ (plus positive TIGRA result, if possible) and normal thorax X-ray assay (normal as absence of any detectable lesion)

Exclusion Criteria:

* Active TB
* Any medical condition or illness that could compromise the volunteer's health if entering the project

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Only a single population is going to be studied: the LTBI, thus people with proof to be M. tuberculosis infected but demonstrating not having active disease.
  As the first approach to demonstrate the Dynamic Hypothesis in humans, up to 6 people will be included as controls.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2009-11; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pere-Joan Cardona, MD, PhD, Study Director — Fundació Institut Germans Trias i Pujol; Cristina Vilaplana, MD, PhD, Principal Investigator — Fundació Institut Germans Trias i Pujol
Locations (3):
- Spain (3):
  - Fundació Institut Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Teknon Foundation, Barcelona

REFERENCES:
- [Background] Cardona PJ. A dynamic reinfection hypothesis of latent tuberculosis infection. Infection. 2009 Apr;37(2):80-6. doi: 10.1007/s15010-008-8087-y. Epub 2009 Mar 23. PMID 19308318
- [Background] Caceres N, Tapia G, Ojanguren I, Altare F, Gil O, Pinto S, Vilaplana C, Cardona PJ. Evolution of foamy macrophages in the pulmonary granulomas of experimental tuberculosis models. Tuberculosis (Edinb). 2009 Mar;89(2):175-82. doi: 10.1016/j.tube.2008.11.001. Epub 2008 Dec 24. PMID 19110471
- [Background] Cardona PJ. New insights on the nature of latent tuberculosis infection and its treatment. Inflamm Allergy Drug Targets. 2007 Mar;6(1):27-39. doi: 10.2174/187152807780077282. PMID 17352686
- [Background] Mack U, Migliori GB, Sester M, Rieder HL, Ehlers S, Goletti D, Bossink A, Magdorf K, Holscher C, Kampmann B, Arend SM, Detjen A, Bothamley G, Zellweger JP, Milburn H, Diel R, Ravn P, Cobelens F, Cardona PJ, Kan B, Solovic I, Duarte R, Cirillo DM; C. Lange; TBNET. LTBI: latent tuberculosis infection or lasting immune responses to M. tuberculosis? A TBNET consensus statement. Eur Respir J. 2009 May;33(5):956-73. doi: 10.1183/09031936.00120908. PMID 19407047
- [Background] Gil O, Diaz I, Vilaplana C, Tapia G, Diaz J, Fort M, Caceres N, Pinto S, Cayla J, Corner L, Domingo M, Cardona PJ. Granuloma encapsulation is a key factor for containing tuberculosis infection in minipigs. PLoS One. 2010 Apr 6;5(4):e10030. doi: 10.1371/journal.pone.0010030. PMID 20386605
- [Background] Cardona PJ. Revisiting the natural history of tuberculosis. The inclusion of constant reinfection, host tolerance, and damage-response frameworks leads to a better understanding of latent infection and its evolution towards active disease. Arch Immunol Ther Exp (Warsz). 2010 Feb;58(1):7-14. doi: 10.1007/s00005-009-0062-5. Epub 2010 Jan 5. PMID 20049645